CLINICAL TRIAL: NCT07324655
Title: The Relationship Between Office Ergonomics, Work Organization, and Musculoskeletal System Complaints Among Medical Secretaries
Brief Title: Association Between Office Ergonomics, Work Organization, and Musculoskeletal Complaints in Medical Secretaries
Status: Not yet recruiting | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH2
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Musculoskeletal Diseases; Ergonomics; Occupational Diseases; Workplace; Pain
Keywords: Medical secretaries; Occupational health; Ergonomics; Musculoskeletal Disease; Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Occupational Diseases; Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Secretaries: Medical secretaries working in hospital settings who are evaluated for office ergonomics, work organization characteristics, and the presence of musculoskeletal complaints using self-reported questionnaires in a single assessment.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study. No intervention is applied. Participants are assessed once using questionnaires to evaluate office ergonomics, work organization, and musculoskeletal complaints.

SUMMARY:
Work-related musculoskeletal complaints are among the most common occupational health issues affecting healthcare staff, especially medical secretaries who spend long hours in sedentary positions and repetitive office tasks. This observational, cross-sectional study aims to investigate the relationship between office ergonomics, work organization, and musculoskeletal system complaints among medical secretaries.

Participants will complete a structured questionnaire that includes demographic and occupational data, ergonomic and work organization characteristics (such as desk and chair setup, posture, computer use, and daily working hours), and self-reported measures of pain and well-being. Postural alignment will be evaluated using the New York Posture Rating Scale (NYPRS), while pain intensity will be assessed with the Visual Analog Scale (VAS). In addition, participants' physical activity level, disability score and stress level will be recorded to examine their potential influence on musculoskeletal symptoms.

The study aims to determine whether poor ergonomic conditions, inadequate posture, low physical activity, and high stress are associated with increased musculoskeletal discomfort, particularly in the neck, shoulders, and lower back regions.

This study is observational and does not include any intervention or experimental treatment. All participation will be voluntary, and data will be collected anonymously. The findings are expected to contribute to preventive strategies and ergonomic improvements to enhance occupational health and comfort among medical secretaries working in healthcare institutions.

DETAILED DESCRIPTION:
Work-related musculoskeletal system disorders are a significant occupational health concern, especially among healthcare professionals performing prolonged sedentary tasks. Medical secretaries are particularly at risk because they spend long hours sitting at a desk, using computers, and performing repetitive upper extremity movements. These conditions may cause pain, postural deviation, and physical or functional limitations that impair quality of life and work efficiency.

This observational, cross-sectional study aims to investigate the relationship between office ergonomics, work organization, and musculoskeletal system complaints among medical secretaries. The study will assess how posture, pain, physical activity, stress, and disability scores interact and contribute to the development of musculoskeletal symptoms.

Participants will include volunteer medical secretaries working in hospital administrative departments. Data will be collected through a structured questionnaire covering demographic and occupational characteristics, ergonomic and organizational factors (e.g., workstation setup, desk and chair suitability, monitor height, working hours, and break frequency), and validated assessment tools.

Postural alignment will be evaluated using the New York Posture Rating Scale (NYPRS), which rates 13 body segments and provides a total score ranging from 13 to 65 points. Pain intensity will be measured by the Visual Analog Scale (VAS). The physical activity level will be assessed using a standardized scale, while stress levels will be measured using a perceived stress questionnaire. Additionally, disability scores will be recorded to evaluate the functional impact of musculoskeletal pain on daily activities and occupational performance.

Statistical analyses will examine correlations between ergonomic conditions, posture, pain, stress, physical activity, and disability scores. Subgroup analyses will explore associations based on age, gender, and years of professional experience.

By identifying key ergonomic and psychosocial risk factors, this study aims to contribute to preventive strategies that improve workplace ergonomics, reduce musculoskeletal discomfort, and enhance the well-being and productivity of medical secretaries in hospital environments.

ELIGIBILITY:
Inclusion Criteria:

* Medical secretaries currently working in a hospital setting
* Aged 18 years or older
* Employed in a desk-based/office position involving computer use
* Working in the current position for at least 6 months
* Presence of self-reported work-related musculoskeletal pain/complaints in at least one body region (e.g., neck, shoulder, upper back, low back, upper extremity) within the last 3 months, assessed by questionnaire
* Willing and able to provide informed consent
* Able to complete self-reported questionnaires

Exclusion Criteria:

* Known spinal deformity or specific spinal disorder (e.g., symptomatic disc herniation/radiculopathy, scoliosis, spondylolisthesis) that could significantly affect musculoskeletal symptoms
* Neurological deficit or neurological disease affecting the musculoskeletal system (e.g., muscle weakness, sensory loss, peripheral neuropathy)
* Diagnosed inflammatory rheumatic disease (e.g., rheumatoid arthritis, ankylosing spondylitis, gout, psoriatic arthritis)
* Major trauma to the neck/upper extremity/spine or orthopedic surgery within the past 6 months
* History of spine surgery (cervical, thoracic, or lumbar)
* Receipt of intensive physical therapy/rehabilitation program or invasive pain procedure (e.g., injection, nerve block) targeting the spine or upper extremity within the past 6 months
* Pregnancy
* Severe cognitive impairment or severe psychiatric disorder that would prevent completion of questionnaires or reliable participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of medical secretaries working in hospital settings who report work-related musculoskeletal pain. Participants are evaluated in a single assessment to examine the association between office ergonomics, work organization characteristics, and musculoskeletal complaints.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence and Severity of Musculoskeletal Complaints | Single assessment (1 day)
  The presence and severity of musculoskeletal complaints among medical secretaries are assessed using a self-reported musculoskeletal questionnaire covering the neck, shoulders, upper back, lower back, and upper extremities, in relation to office ergonomics and work organization factors.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Çelik, Principal Investigator — Ceylanpınar State Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Ceylanpınar State Hospital, Sanliurfa, Ceylanpınar
  - Antalya Training and Research Hospital, Antalya, Muratpaşa

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Durmaz E, Nazlıcan E, Akbaba M.Bir Üniversite Hastanesinde Çalışan Sekreterlerin Üst Ekstremite Kas İskelet Sistemi Yakınmalarının İncelenmesi.Sakarya Tıp Dergisi, 2018, 8(2):432-441
- [Background] Barut Ö, Koçak FA, Kurt EE, Şaş S, Tuncay F, Erdem HR. Sırt veya Bel Ağrısı Olan ve Olmayan Tıbbi Sekreterlerin Omurga Sagittal Eğrilikleri, Fonksiyonel Durum ve Yaşam Kalitesi Düzeylerinin Karşılaştırılması. Harran Üniversitesi Tıp Fakültesi Dergisi. 2020;17(1):91-7.